CLINICAL TRIAL: NCT05923710
Title: Comparison of Primary Anterior Cruciate Ligament Repair With and Without Lateral Extraarticular Tenodesis for Proximal ACL Tears: A Prospective Study
Brief Title: Primary Anterior Cruciate Ligament Repair With and Without Lateral Extraarticular Tenodesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization (Other)
Responsible Party: Principal Investigator, Bulent KARSLIOGLU, Orthopedics and Traumatology specialist,Chief assistant, Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Anterior Cruciate Tear Repair
Record Dates: First submitted 2023-03-23; First posted 2023-06-28 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Anterior Cruciate Ligament Tear
Keywords: proximal anterior cruciate ligament tear; primary repair; Lateral Extraarticular Tenodesis
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Linear Energy Transfer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Primary anterior cruciate ligament repair (Active Comparator): Investigators performed arthroscopic primary repair in 18 patients with proximal ACL tears.
  Interventions: Procedure: Primary anterior cruciate ligament repair; Procedure: Primary anterior cruciate ligament repair and lateral extraarticular tenodesis (LET) with iliotibial band
- Primary anterior cruciate ligament repair and lateral extraarticular tenodesis (LET) (Active Comparator): Investigators performed arthroscopic primary repair and lateral extraarticular tenodesis (LET) with iliotibial band in 20 patients with proximal ACL tears.
  Interventions: Procedure: Primary anterior cruciate ligament repair; Procedure: Primary anterior cruciate ligament repair and lateral extraarticular tenodesis (LET) with iliotibial band

INTERVENTIONS:
Procedure: Primary anterior cruciate ligament repair — Only arthroscopic primary anterior cruciate ligament repair was performed in patients with proximal anterior cruciate ligament tear.
Procedure: Primary anterior cruciate ligament repair and lateral extraarticular tenodesis (LET) with iliotibial band — In addition to primary anterior cruciate ligament repair, lateral extraarticular tenodesis was performed using the iliotibial band.

SUMMARY:
The investigators aimed to compare the clinical results of primary repairs and Lateral Extraarticular Tenodesis applied with primary repairs in the treatment of proximal ACL tears.

DETAILED DESCRIPTION:
The investigators aimed to compare the clinical results of primary repairs and Lateral Extraarticular Tenodesis applied with primary repairs in the treatment of proximal ACL tears.The aim of this study was to determine the potential for improvement with the primary repair of acute ACL tears with the proximal tear, which may be an important advance for improvements in proprioception and preservation of natural kinematics.

ELIGIBILITY:
Inclusion Criteria:

* patients who underwent surgery within the first 3 weeks after injury
* between the ages of 21-40 years,
* attended regular follow-up visits,
* Sherman type 1 proximal ACL tear with relatively preserved synovial sheath
* Sufficient tissue length for re-stretching.

Exclusion Criteria:

* torn ACL in the mid and distal region,
* torn synovial sheath,
* inability to undergo intrasubstance suturing,
* poor tissue quality with retraction,
* multiple ligament injuries and accompanying intra-knee pathologies (meniscal damage, chondral damage),
* previous knee surgery,
* rheumatologic diseases

Ages: 21 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Comparison of functional outcomes between two groups of patients who underwent ACL repair surgery with or without lateral extraarticular tenodesis (LET) with International Knee Documentation Committee (IKDC). | 24 months
  The outcomes were evaluated using various measures, including the International Knee Documentation Committee (IKDC). The IKDC is a patient-completed tool, which contains sections on knee symptoms (7 items), function (2 items), and sports activities (2 items). Scores range from 0 points (lowest level of function or highest level of symptoms) to 100 points (highest level of function and lowest level of symptoms)
Comparison of functional outcomes between two groups of patients who underwent ACL repair surgery with or without lateral extraarticular tenodesis (LET) with Tegner-Lysholm scoring system. | 24 months
  The outcomes were evaluated using various measures, including theTegner-Lysholm scoring system. The Tegner Lysholm scale consists of eight items with each question response being assigned an arbitrary score on an increasing scale. The total score is the sum of each response to the eight questions and may range from 0-100 where higher scores indicate a better outcome with fewer symptoms or disability.

CONTACTS AND LOCATIONS:
Overall Officials: Yasin Guler, Md, Principal Investigator — Metin Sabanci Baltalimani Hospital
Locations (1):
- SBU Prof. Cemil Tascioglu City Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ateschrang A, Schreiner AJ, Ahmad SS, Schroter S, Hirschmann MT, Korner D, Kohl S, Stockle U, Ahrend MD. Improved results of ACL primary repair in one-part tears with intact synovial coverage. Knee Surg Sports Traumatol Arthrosc. 2019 Jan;27(1):37-43. doi: 10.1007/s00167-018-5199-5. Epub 2018 Oct 8. PMID 30298414
- [Result] Abusleme S, Stromback L, Caracciolo G, Zamorano H, Cheyre J, Vergara F, Yanez R. Lateral Extra-articular Tenodesis: A Technique With an Iliotibial Band Strand Without Implants. Arthrosc Tech. 2021 Jan 20;10(1):e85-e89. doi: 10.1016/j.eats.2020.09.029. eCollection 2021 Jan. PMID 33532213
- [Result] Achtnich A, Herbst E, Forkel P, Metzlaff S, Sprenker F, Imhoff AB, Petersen W. Acute Proximal Anterior Cruciate Ligament Tears: Outcomes After Arthroscopic Suture Anchor Repair Versus Anatomic Single-Bundle Reconstruction. Arthroscopy. 2016 Dec;32(12):2562-2569. doi: 10.1016/j.arthro.2016.04.031. Epub 2016 Jun 17. PMID 27324969
- [Result] Anderson MJ, Browning WM 3rd, Urband CE, Kluczynski MA, Bisson LJ. A Systematic Summary of Systematic Reviews on the Topic of the Anterior Cruciate Ligament. Orthop J Sports Med. 2016 Mar 15;4(3):2325967116634074. doi: 10.1177/2325967116634074. eCollection 2016 Mar. PMID 27047983
- [Result] Csintalan RP, Inacio MC, Funahashi TT. Incidence rate of anterior cruciate ligament reconstructions. Perm J. 2008 Summer;12(3):17-21. doi: 10.7812/TPP/07-140. PMID 21331205
- [Result] Di Benedetto P, Di Benedetto E, Fiocchi A, Beltrame A, Causero A. Causes of Failure of Anterior Cruciate Ligament Reconstruction and Revision Surgical Strategies. Knee Surg Relat Res. 2016 Dec 1;28(4):319-324. doi: 10.5792/ksrr.16.007. PMID 27894180
- [Result] DiFelice GS, van der List JP. Clinical Outcomes of Arthroscopic Primary Repair of Proximal Anterior Cruciate Ligament Tears Are Maintained at Mid-term Follow-up. Arthroscopy. 2018 Apr;34(4):1085-1093. doi: 10.1016/j.arthro.2017.10.028. Epub 2018 Jan 17. PMID 29373290
- [Result] DiFelice GS, Villegas C, Taylor S. Anterior Cruciate Ligament Preservation: Early Results of a Novel Arthroscopic Technique for Suture Anchor Primary Anterior Cruciate Ligament Repair. Arthroscopy. 2015 Nov;31(11):2162-71. doi: 10.1016/j.arthro.2015.08.010. PMID 26542201
- [Result] Friden T, Roberts D, Ageberg E, Walden M, Zatterstrom R. Review of knee proprioception and the relation to extremity function after an anterior cruciate ligament rupture. J Orthop Sports Phys Ther. 2001 Oct;31(10):567-76. doi: 10.2519/jospt.2001.31.10.567. PMID 11665744